CLINICAL TRIAL: NCT00934934
Title: Candida in the Respiratory Tract Secretions of Critically Ill Patients and The Efficacy of Antifungal Treatment (The CANTREAT Study): A Prospective, Randomized, Double Blind, Placebo Controlled Pilot Study
Brief Title: Candida in the Respiratory Tract Secretions of Critically Ill Patients and The Efficacy of Antifungal Treatment
Acronym: CANTREAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Daren K. Heyland (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Queen's University (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CANTREAT
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Ventilator Associated Pneumonia; Respiratory Tract Infection
Keywords: Candida; ventilator associated pneumonia; respiratory tract infection; antifungal; biomarker
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Respiratory Tract Infections; Torulopsis | interventions — Saline Solution; Anidulafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline will serve as the placebo solution since the active comparator is clear and colourless.
  Interventions: Other: Normal Saline
- Antifungal (Active Comparator): Patient will receive a dose daily for a total of 14 days
  Interventions: Drug: anidulafungin

INTERVENTIONS:
Other: Normal Saline — Normal Saline
  Arms: Placebo
Drug: anidulafungin — TBA
  Other Names: TBA
  Arms: Antifungal

SUMMARY:
The purpose of the study is to determine whether the effect of treating Candida spp. isolated in the respiratory tract secretions of patients with a clinical suspicion of ventilator associated pneumonia (VAP) on clinical outcomes will be feasible and supported by biomarker data obtained.

DETAILED DESCRIPTION:
Candida spp. is commonly retrieved from microbiologic specimens of ICU patients with suspected VAP. It has been associated with increased systemic inflammation and worse clinical outcomes. This association may be due to the propensity for Candida to colonize those who are sicker, who have increased levels of systemic inflammation and worse clinical outcomes. However, an alternate possibility is that Candida is more than a colonizer and is responsible for the clinical and biochemical features observed. The only way to clarify the pathogenic role of Candida from this patient population is to treat the organism and see if patients improve compared to an untreated group. The purpose of this research program is to conduct such a study to determine if Candida in respiratory tract secretions should be routinely treated in critically ill patients. Since a definitive randomized controlled trial designed to demonstrate a reduction in mortality would be large, require the commitment of large amount of resources including both time and money, the investigators propose to first conduct a small pilot feasibility study.

Eligible patients will be randomized to receive antifungal treatment with anidulafungin or placebo. Following enrollment, study treatment (or placebo) will be started as soon as possible. When the Candida or yeast organisms have been speciated and/or a susceptibility profile is known, the study medication will be adjusted based on susceptibility patterns. The investigators propose to treat with antifungal therapy for a total of 14 days.

Patients will be followed daily for their entire stay in ICU or till day 28, whichever comes first. For patients discharged from the ICU to the ward, they will be followed until study treatment is complete (i.e. day 14). Mortality will be determined for the ICU stay, hospital stay and at 90 days. The investigators will record admission and discharge dates to ICU, step down units, and to hospital.

All patients will have 13 mL of blood/day drawn at baseline, day 3, day 8 and at the end of the treatment period on day 14 (or last day of treatment). The samples will be prepared on site and shipped to a central lab for processing. The investigators will use the blood specimens to measure markers of inflammation (C-reactive protein, Procalcitonin, and Interleukin-6 and others as determined by the investigators), markers of candida presence (b-glucan and other potential future markers) and markers of immune dysfunction (to be determined by investigators).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old)
2. In the ICU > 48 hours
3. Mechanically ventilated (>48 hours)
4. Grow a Candida spp. on respiratory tract secretion culture (either by Bronchoalveolar Lavage or Endotracheal Aspirate) taken on or between 48 hours before or after the day of their suspicion of respiratory tract infection.
5. Develop a clinical suspicion of respiratory tract infection while ventilated as defined by the following criteria (as defined previously in our VAP trial)5:

   * The presence of new, worsening or persistent radiographic features suggestive of pneumonia without another obvious cause AND
   * The presence of any two of the following:

     * Fever > 38C (core temperature)
     * Leukocytosis (>11.0 x109/L) or neutropenia (<3.5 x109/L)
     * Purulent endotracheal aspirates or change in character of aspirates
     * Isolation of pathogenic bacteria from endotracheal aspirates
     * Increasing oxygen requirements

Exclusion Criteria:

1. Patients not expected to be in ICU for more than 72 hours (due to imminent death, withdrawal of aggressive care or discharge).
2. Patients with Candida spp. in the blood or another sterile body site.
3. Patients colonized at other non-pulmonary body site(s) with Candida.
4. Already being treated with antifungal drugs (because of documented fungal infection, pre-emptive therapy, or prophylaxis).
5. Allergy to study drugs (Fluconazole or the Echinocandin on formulary at treating institution).
6. Immunocompromised patients (post-organ transplantation, Acquired Immunodeficiency Syndrome [AIDS], neutropenia [<1000 absolute neutrophils], corticosteroids [>20 mgs/day of prednisone or equivalent for more than 6 months]). These patients are excluded since Candida may be more invasive and these patients are much more likely to require systemic antifungal therapy.
7. Patients with fulminant liver failure or end stage liver disease (Child's Class C).
8. Women who are pregnant or lactating.
9. Enrollment in industry sponsored interventional trial (co-enrollment in other academic studies would be allowed with the proviso that there was no potential interaction between the protocols).
10. Prior randomization in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daren Heyland, MD, Study Chair — Clinical Evaluation Research Unit
Locations (6):
- Canada (6):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital du Sacre-Coeur do Montreal, Montreal, Quebec
  - Hopital l'Enfant-Jesus, Québec

REFERENCES:
- [Background] Safdar N, Dezfulian C, Collard HR, Saint S. Clinical and economic consequences of ventilator-associated pneumonia: a systematic review. Crit Care Med. 2005 Oct;33(10):2184-93. doi: 10.1097/01.ccm.0000181731.53912.d9. PMID 16215368
- [Background] Muscedere JG, Martin CM, Heyland DK. The impact of ventilator-associated pneumonia on the Canadian health care system. J Crit Care. 2008 Mar;23(1):5-10. doi: 10.1016/j.jcrc.2007.11.012. PMID 18359415
- [Background] Van Saene H., Peric M., De La Cal M., Silvestri L.: Pneumonia during Mechanical Ventilation. Anestiologie a Intenzivni Medicina 2004; 15: 89-100.
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Canadian Critical Care Trials Group. A randomized trial of diagnostic techniques for ventilator-associated pneumonia. N Engl J Med. 2006 Dec 21;355(25):2619-30. doi: 10.1056/NEJMoa052904. PMID 17182987
- [Background] Heyland DK, Dodek P, Muscedere J, Day A, Cook D; Canadian Critical Care Trials Group. Randomized trial of combination versus monotherapy for the empiric treatment of suspected ventilator-associated pneumonia. Crit Care Med. 2008 Mar;36(3):737-44. doi: 10.1097/01.CCM.0B013E31816203D6. PMID 18091545
- [Background] Muscedere J, Dodek P, Keenan S, Fowler R, Cook D, Heyland D; VAP Guidelines Committee and the Canadian Critical Care Trials Group. Comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia: prevention. J Crit Care. 2008 Mar;23(1):126-37. doi: 10.1016/j.jcrc.2007.11.014. PMID 18359430
- [Background] Muscedere J, Dodek P, Keenan S, Fowler R, Cook D, Heyland D; VAP Guidelines Committee and the Canadian Critical Care Trials Group. Comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia: diagnosis and treatment. J Crit Care. 2008 Mar;23(1):138-47. doi: 10.1016/j.jcrc.2007.12.008. PMID 18359431
- [Background] Muscedere JG, McColl C, Shorr A, Jiang X, Marshall J, Heyland DK; Canadian Critical Care Trials Group. Determinants of outcome in patients with a clinical suspicion of ventilator-associated pneumonia. J Crit Care. 2008 Mar;23(1):41-9. doi: 10.1016/j.jcrc.2007.12.007. PMID 18359420
- [Background] Rello J, Esandi ME, Diaz E, Mariscal D, Gallego M, Valles J. The role of Candida sp isolated from bronchoscopic samples in nonneutropenic patients. Chest. 1998 Jul;114(1):146-9. doi: 10.1378/chest.114.1.146. PMID 9674461
- [Background] el-Ebiary M, Torres A, Fabregas N, de la Bellacasa JP, Gonzalez J, Ramirez J, del Bano D, Hernandez C, Jimenez de Anta MT. Significance of the isolation of Candida species from respiratory samples in critically ill, non-neutropenic patients. An immediate postmortem histologic study. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):583-90. doi: 10.1164/ajrccm.156.2.9612023. PMID 9279244
- [Background] Senn L, Robinson JO, Schmidt S, Knaup M, Asahi N, Satomura S, Matsuura S, Duvoisin B, Bille J, Calandra T, Marchetti O. 1,3-Beta-D-glucan antigenemia for early diagnosis of invasive fungal infections in neutropenic patients with acute leukemia. Clin Infect Dis. 2008 Mar 15;46(6):878-85. doi: 10.1086/527382. PMID 18260755
- [Background] Odabasi Z, Mattiuzzi G, Estey E, Kantarjian H, Saeki F, Ridge RJ, Ketchum PA, Finkelman MA, Rex JH, Ostrosky-Zeichner L. Beta-D-glucan as a diagnostic adjunct for invasive fungal infections: validation, cutoff development, and performance in patients with acute myelogenous leukemia and myelodysplastic syndrome. Clin Infect Dis. 2004 Jul 15;39(2):199-205. doi: 10.1086/421944. Epub 2004 Jun 28. PMID 15307029
- [Background] Wheeler RT, Fink GR. A drug-sensitive genetic network masks fungi from the immune system. PLoS Pathog. 2006 Apr;2(4):e35. doi: 10.1371/journal.ppat.0020035. Epub 2006 Apr 28. PMID 16652171
- [Background] Azoulay E, Timsit JF, Tafflet M, de Lassence A, Darmon M, Zahar JR, Adrie C, Garrouste-Orgeas M, Cohen Y, Mourvillier B, Schlemmer B; Outcomerea Study Group. Candida colonization of the respiratory tract and subsequent pseudomonas ventilator-associated pneumonia. Chest. 2006 Jan;129(1):110-7. doi: 10.1378/chest.129.1.110. PMID 16424420
- [Background] Delisle MS, Williamson DR, Perreault MM, Albert M, Jiang X, Heyland DK. The clinical significance of Candida colonization of respiratory tract secretions in critically ill patients. J Crit Care. 2008 Mar;23(1):11-7. doi: 10.1016/j.jcrc.2008.01.005. PMID 18359416
- [Background] Heyland et al, WATTCH database. Observational study of the clinical characteristics and biomarker profiles of 569 critically ill patients. Analysis ongoing.
- [Background] Williamson D., Martin A., Perreault M., Delisle M., Muscedere J., Rotstein C., Jiang X., Heyland D. Impact of pulmonary Candida colonization on systemic inflammation in the critically ill. Manuscript in preparation.
- [Background] Magill SS, Swoboda SM, Johnson EA, Merz WG, Pelz RK, Lipsett PA, Hendrix CW. The association between anatomic site of Candida colonization, invasive candidiasis, and mortality in critically ill surgical patients. Diagn Microbiol Infect Dis. 2006 Aug;55(4):293-301. doi: 10.1016/j.diagmicrobio.2006.03.013. Epub 2006 May 15. PMID 16698215
- [Background] Muller V, Viemann D, Schmidt M, Endres N, Ludwig S, Leverkus M, Roth J, Goebeler M. Candida albicans triggers activation of distinct signaling pathways to establish a proinflammatory gene expression program in primary human endothelial cells. J Immunol. 2007 Dec 15;179(12):8435-45. doi: 10.4049/jimmunol.179.12.8435. PMID 18056390
- [Background] Inoue K, Takano H, Oda T, Yanagisawa R, Tamura H, Ohno N, Adachi Y, Ishibashi K, Yoshikawa T. Candida soluble cell wall beta-D-glucan induces lung inflammation in mice. Int J Immunopathol Pharmacol. 2007 Jul-Sep;20(3):499-508. doi: 10.1177/039463200702000308. PMID 17880763
- [Background] Sakurai T, Ohno N, Yadomae T. Effects of fungal beta-glucan and interferon-gamma on the secretory functions of murine alveolar macrophages. J Leukoc Biol. 1996 Jul;60(1):118-24. PMID 8699115
- [Background] Nseir S, Jozefowicz E, Cavestri B, Sendid B, Di Pompeo C, Dewavrin F, Favory R, Roussel-Delvallez M, Durocher A. Impact of antifungal treatment on Candida-Pseudomonas interaction: a preliminary retrospective case-control study. Intensive Care Med. 2007 Jan;33(1):137-42. doi: 10.1007/s00134-006-0422-0. Epub 2006 Nov 8. PMID 17115135
- [Background] Tschaikowsky K, Hedwig-Geissing M, Schiele A, Bremer F, Schywalsky M, Schuttler J. Coincidence of pro- and anti-inflammatory responses in the early phase of severe sepsis: Longitudinal study of mononuclear histocompatibility leukocyte antigen-DR expression, procalcitonin, C-reactive protein, and changes in T-cell subsets in septic and postoperative patients. Crit Care Med. 2002 May;30(5):1015-23. doi: 10.1097/00003246-200205000-00010. PMID 12006796
- [Background] Williamson D., Albert M., Perreault M., Delisle M., Muscedere J., Rotstein C.Jiang X., Day A. ,Heyland D. Effect of Candida spp. in respiratory tract secretions on systemic inflammation. Submitted to SCCM for Feb. 2009
- [Background] Presterl E, Lassnigg A, Mueller-Uri P, El-Menyawi I, Graninger W. Cytokines in sepsis due to Candida albicans and in bacterial sepsis. Eur Cytokine Netw. 1999 Sep;10(3):423-30. PMID 10477399
- [Background] Christofilopoulou S, Charvalos E, Petrikkos G. Could procalcitonin be a predictive biological marker in systemic fungal infections?. Study of 14 cases. Eur J Intern Med. 2002 Dec;13(8):493-495. doi: 10.1016/s0953-6205(02)00160-7. PMID 12446193
- [Background] Reade MC, Angus DC. The clinical research enterprise in critical care: what's right, what's wrong, and what's ahead? Crit Care Med. 2009 Jan;37(1 Suppl):S1-9. doi: 10.1097/CCM.0b013e318192074c. PMID 19104206
- [Background] van Teijlingen E, Hundley V. The importance of pilot studies. Nurs Stand. 2002 Jun 19-25;16(40):33-6. doi: 10.7748/ns2002.06.16.40.33.c3214. PMID 12216297
- [Background] Arnold DM, Burns KE, Adhikari NK, Kho ME, Meade MO, Cook DJ; McMaster Critical Care Interest Group. The design and interpretation of pilot trials in clinical research in critical care. Crit Care Med. 2009 Jan;37(1 Suppl):S69-74. doi: 10.1097/CCM.0b013e3181920e33. PMID 19104228
- [Background] Canadian Institutes of Health Research. Available at: www.cihr.ca Accessed February 9, 2009.
- [Derived] Albert M, Williamson D, Muscedere J, Lauzier F, Rotstein C, Kanji S, Jiang X, Hall M, Heyland D. Candida in the respiratory tract secretions of critically ill patients and the impact of antifungal treatment: a randomized placebo controlled pilot trial (CANTREAT study). Intensive Care Med. 2014 Sep;40(9):1313-22. doi: 10.1007/s00134-014-3352-2. Epub 2014 Jul 1. PMID 24981955
- [Derived] Williamson DR, Albert M, Perreault MM, Delisle MS, Muscedere J, Rotstein C, Jiang X, Heyland DK. The relationship between Candida species cultured from the respiratory tract and systemic inflammation in critically ill patients with ventilator-associated pneumonia. Can J Anaesth. 2011 Mar;58(3):275-84. doi: 10.1007/s12630-010-9439-5. Epub 2010 Dec 14. PMID 21287306

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One pt was mistakenly randomized to intervention without Candida, so was moved to observational group prior to starting treatment
Period: Overall Study
Arm/Group | Placebo | Antifungal
Started | 30 | 31
Completed | 29 | 31
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Antifungal | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (13.8) | 57.6 (17.1) | 60.3 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Recruitment Rate
Description: Overall recruitment rate per site
Time Frame: 32 months
Population: This outcome measure was pre-specified to be for overall participants not by group. It was a reflection of how recruitment went for this protocol overall not by group.
Measure: Number; unit: participants per site /month
Units Other Than Participants: sites
Arm/Group | Overall
Number analyzed (Participants) | 61
Number analyzed (sites) | 5
participants per site /month | 0.6

2. Secondary Outcome: Duration of Stay in ICU
Description: Measure of the duration of participant stay in the ICU
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
days | 11.5 [8 to 20] | 13 [8 to 28]

3. Secondary Outcome: Ventilator Free Days
Description: Number of days in ICU free of ventilation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
days | 8 [6 to 11] | 9 [4 to 10]

4. Secondary Outcome: ICU Free Days
Description: Number of days free of ICU
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
days | 14 [0 to 17] | 4 [0 to 17]

5. Secondary Outcome: Antibiotic Free Days 28-day Post Randomization
Description: Number of days free of antibiotic use within the first 28 days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
days | 16 [12 to 20] | 10 [0 to 20]

6. Secondary Outcome: Hospital Length of Stay
Description: Measure of the duration of the participant's hospital stay
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
days | 29 [17 to 38] | 28 [18 to 46]

7. Secondary Outcome: (SOFA) Post Randomization
Description: Sequential organ failure assessment. 0-24 The higher the number the more severe organ failure
Time Frame: post randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Antifungal
Number analyzed (Participants) | 29 | 31
score on a scale | 5.9 (3.3) | 5.9 (3.6)

8. Secondary Outcome: Sequential Procalcitonin
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | VAP withCandida | VAP Without Candida
Number analyzed (Participants) | 56 | 21
ng/ml | 3.0 (8.8) | 22.5 (89.4)

9. Secondary Outcome: C-reactive Protein
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | VAP withCandida | VAP Without Candida
Number analyzed (Participants) | 56 | 21
mg/l | 133 (115) | 145.7 (104)

10. Secondary Outcome: Interleukin-6
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | VAP withCandida | VAP Without Candida
Number analyzed (Participants) | 56 | 21
pg/ml | 97.5 (183) | 3 (10.3)

11. Secondary Outcome: B-glucan Levels
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | VAP withCandida | VAP Without Candida
Number analyzed (Participants) | 56 | 21
pg/ml | 116 (171) | 129.1 (190.5)

ADVERSE EVENTS:
Description: "0" Total Number of Participants at Risk (e.g.., serious and other [non-serious] adverse events were not collected or assessed as part of the study).
Arm/Group | Placebo | Antifungal
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We had an overall enrolment rate/month of 0.6 patients/site for the randomized trial. Consequently, recruitment was halted prematurely despite efforts to optimize enrolment because of difficulty in recruiting patients and diminishing study resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No